CLINICAL TRIAL: NCT03020550
Title: Physiologic and Behavioral Correlates of GERD Symptom Severity
Brief Title: Correlates of GERD Symptom Severity
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Michelle Dossett, MD, PhD, MPH, Assistant Physician, Massachusetts General Hospital
Other Study IDs: 2016P001628; 1K23AT009218 (NIH)
Record Dates: First submitted 2016-12-20; First posted 2017-01-13 (Estimated); Results first posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-12

CONDITIONS: GERD
Keywords: GERD; Galvanic Skin Response; Heart Rate Variability
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GERD Patients: Subjects with active GERD symptoms.

SUMMARY:
This is a pilot study measuring physiologic and behavioral correlates of symptom severity in adult patients with gastroesophageal reflux disease (GERD).

DETAILED DESCRIPTION:
Subjects will complete questionnaires regarding their GERD-related symptoms and have a visit with a study clinician regarding their symptoms. We will measure heart rate variability and galvanic skin response in patients during the visits and video record the visits. Subjects will complete a daily GERD symptom diary for 2 weeks and then return to the study center to complete additional questionnaires and an exit interview.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 21-70 years old
* Heartburn symptoms 3 or more days per week with an average daily symptom severity of 3 or more on a 7 day baseline symptom diary
* English language proficiency
* Willingness to be videotaped and connected to physiologic monitoring devices during the visit

Exclusion Criteria:

* Diagnosis of Crohn's disease, systemic sclerosis, known active ulcer disease, gastric cancer, or untreated/active Barrett's esophagitis based on subject self-report and/or medical record review
* Heavy alcohol use (> 6 drinks/week for women and > 13 drinks/week for men)
* Pregnant women.
* Dementia or significant memory difficulties
* Severe, unstable psychiatric disease
* Greater than 15 doses of nonsteroidal anti-inflammatory drugs (NSAIDS) within the prior 30 days (aspirin ≤ 325 mg daily permitted) or ongoing NSAID use at a level deemed likely to interfere with the study
* Failure to complete the baseline symptom diary for at least 6 of 7 days
* Change in GERD treatment regimen within the last 2 weeks (subjects may use antacids, H2 receptor blockers, and/or proton pump inhibitors as long as they are symptomatic on a stable regimen)
* Allergy to adhesives
* Inability to provide informed consent

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with active GERD-related symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Dossett, MD, PHD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Visit: A standardized visit (based on a pre-set question template) modeled after a primary care visit focused on evaluating GERD symptoms.
- Expanded Visit: A standardized visit (based on a pre-set question template) modeled after an integrative medicine visit for GERD symptoms. The Expanded Visit includes all of the questions in the Standard Visit plus additional questions about the nature of the GI symptoms (e.g., taste of reflux, food cravings and aversions), other health issues, and the patient's temperament (e.g., shy, anxious, caring). Some of these questions address the patient's "constitutional type" as might be assessed by some integrative practitioners (e.g., tell me about your sleep; do you tend to be hot or cold?).
Period: Overall Study
Arm/Group | Standard Visit | Expanded Visit
Started | 8 | 16
Completed | 8 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Visit: Patients with GERD receiving a standard medical visit
- Expanded Visit: Patients with GERD receiving an expanded medical visit modeled after an integrative medicine consultation
- Total: Total of all reporting groups
Arm/Group | Standard Visit | Expanded Visit | Total
Number analyzed (Participants) | 8 | 16 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (15.7) | 41.1 (16.7) | 39.9 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 13 | 18
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 16 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 7 | 10 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 16 | 24
Average Daily GERD Symptom Severity [Mean (Standard Deviation); unit: units on a scale] — Severity of GERD symptoms were assessed by participant self-report on a 7-day symptom diary for one week immediately prior to enrolling in the study. Possible daily scores ranged from 0-12 with higher scores indicating more severe symptoms (sum of daytime heartburn, nighttime heartburn, and acid regurgitation symptoms each rated 0-4 in severity [none, mild, moderate, severe, very severe]). Daily values across each of the 7 days were averaged to create the average daily GERD symptom severity score. Adapted from: Miner P, et. al. Am J Gastroenterol. 2002 Jun;97(6):1332-1339. PMID: 12094846
  units on a scale | 3.90 (1.7) | 2.95 (1.2) | 3.26 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Association of Change in Patient's GSR From Beginning to End of Study Visit With GERD Symptom Severity 2 Weeks Later
Description: Galvanic skin response (GSR) was measured with a device from ADInstruments during the baseline study visit. Values ranged from 0.93 - 12 micro-Siemens (μS). Change in GSR was calculated as mean value of GSR for the first 2 minutes of the study visit minus mean value of GSR for the last 2 minutes of the study visit.
Time Frame: Beginning to end of study visit (1 hour or less for change in GSR)
Population: Intent to treat analysis. Subjects with missing GSR data (due to equipment malfunction) were not included in the final analysis.
Measure: Mean (Standard Deviation); unit: micro-Siemens
Arm/Group | Standard Visit | Expanded Visit
Number analyzed (Participants) | 7 | 9
micro-Siemens | -0.94 (1.3) | -1.70 (1.1)
Statistical Analysis 1: Comparison: Standard Visit vs Expanded Visit; The outcome measure was calculated using a general linear model with average daily post GERD symptom severity as the dependent variable with the following independent variables: baseline average GERD symptom severity and change in GSR (galvanic skin response). No term for visit type assignment was included in the model; Test type: Superiority; p = 0.034, ANOVA; Adjusted for baseline GERD symptom severity

2. Primary Outcome: Association of Change in Patient's High Frequency HRV From Beginning to End of Study Visit With GERD Symptom Severity 2 Weeks Later
Description: Heart rate variability (HRV) was measured using a device from ADInstruments gathering data at 256 Hz. We used the RMSSD (Root Mean Square of the Successive Differences) value as a proxy for high frequency HRV. Measured values ranged from 0 - 150 msec. Change in high frequency HRV was calculated as the RMSSD value for the first 5 minutes of the study visit minus the RMSSD value for the last 5 minutes of the study visit.
Time Frame: Beginning to end of study visit (1 hour or less for change in HRV/RMSSD)
Population: Intent to treat analysis.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Standard Visit | Expanded Visit
Number analyzed (Participants) | 8 | 16
milliseconds | -0.26 (8.3) | 2.5 (10.3)
Statistical Analysis 1: Comparison: Standard Visit vs Expanded Visit; The outcome measure was calculated using a general linear model with average daily post GERD symptom severity as the dependent variable with the following independent variables: baseline average GERD symptom severity and change in RMSSD (high frequency HRV). No term for visit type assignment was included in the model; Test type: Superiority; p = 0.56, ANOVA; Adjusted for baseline GERD symptom severity

3. Primary Outcome: Correlation Between Concordance in GSR Between Patient and Physician During the Study Visit and Percent Change in Patients' GERD Symptoms Over 2 Weeks
Description: Concordance in galvanic skin response (GSR) between patient and physician was calculated using an established approach (Marci CD, 2007; PMID 17299296) to create a single index value for the visit. The natural logarithm of this value was taken to reduce skew. A value greater than 0 means more than 50% concordance in the data, a value less than zero means less than 50% concordance in the data.
Time Frame: Beginning to end of study visit (1 hour or less for concordance between patient and physician GSR)
Population: Intent to treat. Subjects with missing GSR data (due to equipment malfunction) were not included in the final analysis.
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Standard Visit | Expanded Visit
Number analyzed (Participants) | 7 | 9
Index | -0.0536 (0.19) | 0.199 (0.38)
Statistical Analysis 1: Comparison: Standard Visit vs Expanded Visit; The outcome measure was calculated using a Pearson correlation to compare the session index representing the amount of concordance in GSR between patient and physician and the percent change in patients' GERD symptoms. Visit type assignment was not included in the analysis; Test type: Superiority; p = 0.80, Pearson's correlation test

4. Other Pre Specified Outcome: Post GERD Symptom Severity
Description: GERD symptom severity at follow-up was assessed by self-report on a 7-day symptom diary (symptoms collected days 8-14 after the study visit). Possible daily scores ranged from 0-12 with higher scores indicating more severe symptoms (sum of daytime heartburn, nighttime heartburn, and acid regurgitation symptoms each rated 0-4 in severity [none, mild, moderate, severe, very severe]). Daily scores across the 7 days were averaged to create the Post GERD symptom severity score. Adapted from: Miner P, et. al. Am J Gastroenterol. 2002. PMID: 12094846.
Time Frame: 2 weeks (baseline and 2 week follow-up)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Visit | Expanded Visit
Number analyzed (Participants) | 8 | 16
score on a scale | 3.77 (1.48) | 2.41 (1.67)

5. Other Pre Specified Outcome: Percent Change in Patient's GERD Symptoms
Description: Percent change in patient's GERD symptoms was calculated as: (post GERD symptom severity - baseline GERD symptom severity) / baseline GERD symptom severity*100.
  GERD symptom severity scores were averaged across 7 day baseline and follow-up periods from a symptom diary (adapted from Miner P, 2002; PMID 12094846). Scores ranged from 0-12 with higher scores indicating more severe symptoms (sum of daytime heartburn, nighttime heartburn, and acid regurgitation each rated 0-4 in severity [none, mild, moderate, severe, very severe]).
Time Frame: 2 weeks (baseline and 2 week follow-up)
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Standard Visit | Expanded Visit
Number analyzed (Participants) | 8 | 16
Percent change | 10.3 (45) | -12.2 (58)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Standard Visit | Expanded Visit
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/16
Other Adverse Events (participants affected / at risk) | 1/8 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Visit (N=8) | Expanded Visit (N=16)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — 1 subject developed gastroenteritis and presented to the emergency department where they received IV fluids. Adverse event deemed not related to the study intervention.

LIMITATIONS AND CAVEATS:
Equipment malfunction led to incomplete data collection for some subjects, reducing the total number of subjects in some of the data analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT03020550/Prot_SAP_000.pdf